CLINICAL TRIAL: NCT04884698
Title: "Electromagnetical Stimulation of the Phrenic Nerve to Generate Contraction of the Diaphragm in Healthy Subjects and Anaesthetized and Intubated Patients - a Feasibility Study"
Brief Title: "Electromagnetical Stimulation of Phrenic Nerve to Generate Contraction of the Diaphragm"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stimit AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Stimit swiss I
Record Dates: First submitted 2021-04-30; First posted 2021-05-13 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-06

CONDITIONS: Healthy Subjects; Elective Surgical Procedure

STUDY DESIGN:
Intervention Model Description: Open-label, sponsor-initiated feasibility study. 2 groups of patients treated - healthy subjects and elective surgery patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phrenic nerve stimulation with Stimit Activator (Experimental)
  Interventions: Device: Stimit Activator

INTERVENTIONS:
Device: Stimit Activator — The Stimit Activator Device is composed of three components.
  1. A magnetic stimulator generating current pulses
  2. A novel Stimit coil design optimized for phrenic nerve stimulation
  3. A coil positioning device for quick, easy and reproducible coil positioning

SUMMARY:
The scientific study is intended to show that external non-invasive electromagnetic stimulation can be used to safely and effectively stimulate the phrenic nerve in awake healthy subjects as well as in ventilated, anesthetized patients and that the stimulation can generate a diaphragmatic contraction that generates significant breath volume - a Controlled Own Breath (COB).

Also of interest is the reproducibility of the generated diaphragmatic movements and the reliability of different feedback signals for detecting the generated diaphragmatic contraction. This applies to inspiration and expiration detection for subsequent synchronization mechanisms of the magnetic stimulator for patient-initiated breathing as well as to contraction intensity. Further, the characterization of the position finding process is of great importance, so that technical developments can further simplify the process of coil positioning in the future. The possible occurrence of discomfort and pain sensation will also be investigated in awake healthy volunteers. Different stimulation protocols will be used.

Finally, it will be investigated whether an adjusted coil position still triggers reproducible diaphragmatic contractions after removal and repositioning in the same configuration. The knowledge gained will be used to further develop the technique and to prepare a study in critically ill, ventilated patients where the diaphragmatic muscle is to be treated preventively by stimulating the phrenic nerve, in order to prevent atrophy of the muscle.

ELIGIBILITY:
Inclusion Criteria:

* Persons aged > 18 years
* Applicable for Group 2: planned for elective surgery
* No relevant pre-existing conditions - corresponding to American Society of Anesthesiologists (ASA) level of I-II.
* Written informed consent by the patient for participation in the study given

Exclusion Criteria:

* chronic lung diseases (bronchial asthma, COPD)
* known diaphragmatic weakness
* known neurological conditions with motor muscle weakness
* known paralysis of the phrenic nerve
* conditions that limit the mobility of the diaphragm (high intra-abdominal pressure, ascites, BMI >30)
* not able to read and understand the national language German
* skin lesions, infections or strictures in the neck area
* persons with Implanted cardiac support systems (pacemaker, implanted defibrillator)
* persons with implanted medical pumps
* pregnant women
* persons deprived of liberty by administrative or judicial decision or under legal guardianship.
* Participation in another clinical trial
* Applicable for group 2 (intubated and mechanically ventilated) patients: Exclusion criteria at the time of stimulation:

  * Unstable patient after induction of anesthesia and intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Change in airway pressure / endpoint Group 1: | During stimulation
  The primary outcome / endpoint is the change in airway pressure at the mouth during stimulation as seen with or without the use of the ventilator
Discomfort / pain during stimulation measured by Visual Analogue Scale / endpoint Group 1: | During stimulation
  The primary outcome / endpoint is the level of discomfort / pain during stimulation, measured by Visual Analogue Scale(0-100, with 100 being worst pain / discomfort)
Change in airway pressure / endpoint Group 2: | During stimulation
  The primary outcome / endpoint is the change in airway pressure during stimulation as seen with or without the use of the ventilator during stimulation.

SECONDARY OUTCOMES:
Diaphragmatic contraction | During stimulation
  Diaphragmatic contraction at 20 percent / 30 percent / 40 percent stimulation intensity at the optimal stimulation site, at 25 Hz and 2s stimulation time
Feedback signals | During stimulation
  Change of the maximum value of the feedback signals in percent of the maximum depending on the coil position (in 0.5 cm steps; at least 3 steps in each direction)
Time stimulation start to end | During stimulation
  Time (mean value & standard deviation) between stimulation start and stimulation end (trigger signal start and end) until the feedback signals from:
  * the abdominal belt,
  * the Diaphragm Thickening Fraction ((TFdi) according to standard procedure, measured via ultrasound during stimulation), and
  * the Diaphragm Excursion Signal "respons" (measured by ultrasound during stimulation)
Correlation stimulation intensity and diaphragm contraction | During stimulation
  Correlation between stimulation intensity (power output in percent) and diaphragm contraction, measured by tidal volume, at the optimal coil position at given frequency (25 Hz) and given stimulation duration
Optimal stimulation site - distance | During stimulation
  Distance from anatomical landmark (a) to optimal stimulation site (b) and phrenic nerve (c) using ultrasound and between b and c
Optimal stimulation site - time | During stimulation
  Time from the start of coil positioning to finding a coil positioning which produces the maximum diaphragmatic contraction at a given stimulation intensity and frequency of 25 Hz
Tidal volumes | During stimulation
  The mean and standard deviation of generated tidal volumes for ten stimulations performed without the subject being ventilated
Skin reactions / musle activation | During stimulation
  For Group 1: evaluation of stimulation-induced local skin reactions or muscle activation leading to paresthesia in the dental area
Safety outcome | During stimulation and postoperatively, usually within 2-3 hours
  The safety outcome/ endpoint is the occurrence of the following events during stimulation:
  * Device related Adverse Events
  * Device related Serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Michael Baumberger, MD, Principal Investigator — Swiss Paraplegic Center Nottwil
Locations (1):
- Swiss Paraplegic centre, Nottwil, Switzerland

IPD SHARING:
Plan to Share IPD: No